CLINICAL TRIAL: NCT04124991
Title: A Single-arm, Open-label, Safety and Efficacy Study of Radioembolization With Yttrium-90 Microspheres in Combination With Durvalumab (MEDI4736) in Locally Advanced and Unresectable Hepatocellular Carcinoma (HCC) (SOLID)
Brief Title: Safety and Efficacy Study of Radioembolization in Combination With Durvalumab in Locally Advanced and Unresectable HCC
Acronym: SOLID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yoon Jun Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLID
Record Dates: First submitted 2019-08-20; First posted 2019-10-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Durvalumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Transarterial radioembolization (TARE) with yttrium-90 microspheres will be employed in combination with an intravenous (IV) dose of 1500 mg durvalumab every 4 weeks (Q4W) until PD. TARE will be performed 1-2 weeks (7 to 14 days) before the first dose of durvalumab and a maximum of 2 more times during the treatment period, per Investigator discretion. If additional TARE is performed, the interval between additional TARE treatments and administration of durvalumab should be at least 1 week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Yttrium-90 Microspheres in Combination with Durvalumab (Experimental): Transarterial radioembolization (TARE) with yttrium-90 microspheres will be employed in combination with an intravenous (IV) dose of 1500 mg durvalumab every 4 weeks (Q4W) until PD. TARE will be performed 1-2 weeks (7 to 14 days) before the first dose of durvalumab and a maximum of 2 more times during the treatment period, per Investigator discretion. If additional TARE is performed, the interval between additional TARE treatments and administration of durvalumab should be at least 1 week.
  Interventions: Drug: Durvalumab; Radiation: Radioembolization

INTERVENTIONS:
Drug: Durvalumab — Radioembolization with Yttrium-90 Microspheres
  Other Names: Imfinzi®
Radiation: Radioembolization — Radioembolization with Yttrium-90 Microspheres
  Other Names: TheraSphere™

SUMMARY:
Safety and Efficacy Study of Radioembolization with Yttrium-90 Microspheres in Combination with Durvalumab in Locally Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
This is a single arm, open-label study to evaluate safety and efficacy of Radioembolization with Yttrium-90 Microspheres in Combination with Durvalumab in Locally Advanced and Unresectable Hepatocellular Carcinoma which to be implemented at a single site in Korea.

Transarterial radioembolization (TARE) with yttrium-90 microspheres will be employed in combination with an intravenous (IV) durvalumab until PD. TARE will be performed before the first dose of durvalumab. Exploratory biomarker testing will be done on tumor tissues prior to treatment and plasma samples prior to treatment and at the time of PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unequivocal HCC confirmed histologically or diagnosed radiologically
* Locally advanced HCC
* Must have at least 1 untreated measurable disease
* Child-Pugh score ≤7 points
* Adequate normal organ and marrow function.

Exclusion Criteria:

* Eligible for potentially curative treatment (surgical resection, radio-frequency ablation or immediate liver transplantation)
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti- Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody
* Any other concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, papillary thyroid cancer, early gastric cancer, or other cancer for which the patient has been disease-free for at least five years.
* Evidence of extrahepatic metastasi(e)s, except for regional lymph node(s) involvement
* History of leptomeningeal carcinomatosis , History of active primary immunodeficiency
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.

Exclusion Criteria Specific to Radioembolization:

•The screening angiogram and technetium-99m macroaggregated albumin (99mTc-MAA) scan are used to determine lobar liver volume from CT or MR images, to identify vascular shunting to the GI tract requiring use of angiographic occlusion techniques and to determine the lung shunt fraction.

Patients who are ineligible to radioembolization meeting the following criteria will not be included in the study. Additional patients will be screened to replace those patients.

* Deposition of yttrium-90 microspheres to the GI tract that cannot be corrected by placement of the catheter distal to collateral vessels or the application of standard angiographic techniques, such as coil embolization to prevent deposition of yttrium-90 microspheres in the GI tract.
* Exposure of radiation to the lungs exceeds 30 Gray (Gy) for a single infusion or 50 Gy cumulative for all infusions of yttrium-90 microspheres.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
TTP | From date of enrollment until the date of first documented progression, assessed up to 12 months
  to evaluate time to progression (TTP) from enrolment using Modified Response Evaluation Criteria in Solid Tumors (mRECIST).

SECONDARY OUTCOMES:
OS | From date of enrollment until the date of first documented progression, assessed up to 12 months
  Overall Survival (OS) from first dose of study drug until the time of data cut-off, as determined by the Investigator.
ORR | From date of enrollment until the date of first documented progression, assessed every 8 weeks up to 12 months.
  Objective Response Rate (ORR) of Target Lesion(s) and Non-Target Lesion(s)
Number of participants with treatment-related adverse events | Until 30 days after radioembolization with yttrium-90 microspheres or the last dose of durvalumab
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jun Kim, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No